CLINICAL TRIAL: NCT03886636
Title: The Effectiveness of Neuroscience Pain Education Combining Manual Therapy in Patients with Chronic Low Back Pain: a Single-blinded Randomized Controlled Trial
Brief Title: Neuroscience Pain Education in Patients with Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ismail Saracoglu, Principle Investigator, Kutahya Health Sciences University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: KutahyaMSU
Record Dates: First submitted 2019-03-19; First posted 2019-03-22 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2019-03

CONDITIONS: Chronic Low Back Pain; Manual Therapy; Neuroscience Pain Education
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Neuroscience pain education group (Experimental): in Group 1, participants received Neuroscience pain education, manual therapy and a home exercise program.
  Interventions: Other: neuroscience pain education; Other: manual therapy; Other: home exercises
- Manual therapy group (Experimental): in Group 2, participants received manual therapy and a home exercise program.
  Interventions: Other: manual therapy; Other: home exercises
- Control group (Active Comparator): in Group 3, participants received home exercise program only.
  Interventions: Other: home exercises

INTERVENTIONS:
Other: neuroscience pain education — A total of 4 NPE (Neuroscience paine education) sessions were held, once each week, before an MT session. The NPE sessions were conducted by an experienced physiotherapist certified in NPE in face-to-face, one-on-one sessions lasting 40-45 minutes. In NPE, the patient is taught about the physiology of pain, central sensitization, representation of the different body regions in the brain, pain-related changes in body perception, and the psychosocial dimensions of pain.
  Arms: Neuroscience pain education group
Other: manual therapy — In our study, Manual therapy (MT) was individualized according to each patient's response to treatment. In this method, the physiotherapist identifies and performs techniques suitable for the patient's symptoms. If the selected techniques do not have a direct positive effect on the patient's symptoms, they are replaced with other techniques.MT were performed in a total of 8 sessions, held twice a week for 4 weeks. Treatment sessions lasted an average of 40-45 minute.The entire treatment program was carried out by the same physiotherapist who is trained and experienced in this area.
  Arms: Manual therapy group; Neuroscience pain education group
Other: home exercises — All participants in all groups were assigned the home exercise program. The program aims to increase strength and flexibility of the abdominal, erector spinae, gluteal, quadriceps, and hamstring muscles. The participants were then asked to perform all of the exercises with 10 repetitions of each exercise 3 times a day for 4 weeks.

SUMMARY:
The cognitive educational strategies such as neuroscience pain education, has been a popular and promising technique for treatment patients with chronic pain. However, there are not sufficient randomized controlled and blinded studies to explore clinical effectiveness of these techniques. Therefore, the aim of this study was determining the short- and mid-term effects of neuroscience pain education combined with manual therapy and home exercise on pain level, disability, and kinesiophobia in patients with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Volunteered to participate in the study.
* Patients with 18-65 years
* Had low back pain for at least 6 months,
* Reported pain severity of 5 or greater according to the numeric pain rating scale
* Used pregabalin and gabapentin derivatives,

Exclusion Criteria:

* Previous spine or lower extremity surgery
* Severe osteoporosis
* Spondyloarthropathy
* Spondylolisthesis
* Lumbar stenosis
* Systemic inflammatory diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale (NPRS) | Change from Baseline NPRS at 4th weeks and 12th weeks
  The NPRS was used to assess the participants' pain levels. In the NPRS, patients are asked to verbally rate the severity of their pain on a scale from 0 to 10. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | Change from Baseline ODI at 4th weeks and 12th weeks
  The participants' level of functioning was evaluated using the Turkish adaptation of the ODI. The scale comprises 10 items, each with 6 options worth 0 to 5 points. For each item, participants are asked to mark the option that best describes their current condition. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Back Performance Scale (BPS) | Change from Baseline BPS at 4th weeks and 12th weeks
  The BPS includes five tests of trunk mobility. Each test is scored from 0 to 3 based on the observed level of physical performance, and total score ranges from 0 to 15 points (18). High score indicates poor performance.
Tampa Scale for Kinesiophobia (TSK) | Change from Baseline TSK at 4th weeks and 12th weeks
  TSK was used for the assessment of kinesiophobia. The items are rated on a 4-point Likert-type scale (1=definitely disagree, 4=completely agree) and the total score is between 17 and 68 points. Higher total score indicates higher level of kinesiophobia.

CONTACTS AND LOCATIONS:
Locations (1):
- Yoncali Physical Therapy and Rehabilitation Hospital, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No